CLINICAL TRIAL: NCT00000933
Title: Effects of Prophylaxis for Disseminated Mycobacterium Avium Complex (MAC) Disease With Azithromycin Versus Deferred Prophylaxis on Carriage of Antibiotic-Resistant Streptococcus Pneumoniae: A Substudy of the CR-MAC Protocol (CPCRA 048)
Brief Title: Effects of MAC Preventive Therapy on Disease-Causing Bacteria in HIV-Infected Patients: A Substudy of CPCRA 048
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 054; 11607 (Registry Identifier: DAIDS ES); Parent Study CPCRA 048
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections; Pneumococcal Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Antibiotics, Macrolide; Azithromycin; Drug Administration Schedule; Drug Resistance, Microbial; Carrier State; Streptococcus pneumoniae
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Pneumococcal Infections; AIDS-Related Opportunistic Infections

SUMMARY:
Some people who have taken azithromycin to prevent MAC (Mycobacterium avium Complex, a bacterial infection common in HIV-infected persons) have been found to carry antibiotic-resistant bacteria (germs that grow despite the presence of drugs used to kill them). The purpose of this study is to see if people who take azithromycin carry more antibiotic-resistant bacteria than people who have chosen to delay MAC preventive therapy.

When bacteria like Streptococcus (a type of bacteria that causes pneumonia and meningitis) are frequently exposed to antibiotics, the bacteria can become resistant to the drugs. MAC preventive therapy uses antibiotics, but this can make it difficult to treat other infections caused by bacteria that have become resistant in HIV-infected persons. If MAC preventive therapy is delayed, Streptococcus in the body may be less likely to develop resistance. Therefore, if the patient does get a Streptococcus infection, it will be easier to treat because it is not resistant to the antibiotics.

DETAILED DESCRIPTION:
Streptococcus pneumoniae is a leading cause of bacteremia, pneumonia, meningitis, and otitis media in the United States. Prior to 1987, this organism was uniformly susceptible to penicillin; since then, however, increasing numbers of isolates resistant to penicillin, as well as to other common antibiotics, have been identified. Frequent exposure to antibiotics has been documented as an important risk factor for the emergence of resistant organisms in HIV-infected patients, who are more likely than uninfected people to be colonized with antibiotic-resistant strains of S. pneumoniae. This substudy is the first to examine the effects of withdrawing or delaying the initiation of prophylaxis (in this case, MAC prophylaxis) on the prevalence of antibiotic-resistant pneumococci in a prospective manner.

Study participants are a subset of those enrolled in the CR-MAC Protocol (CPCRA 048). Oropharyngeal swabs are taken at baseline and 4 months after randomization, and are used to isolate S. pneumoniae in culture. These isolates are tested for susceptibility to macrolides, penicillin, cephalosporins, quinolones, and TMP-SMX. The rates of pneumococcal colonization at baseline and 4 months after randomization are determined and used to estimate the impact of deferring MAC prophylaxis on carriage of antibiotic-resistant S. pneumoniae.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are enrolled in CPCRA 048.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: El-Sadr W, Study Chair; Burman W, Study Chair
Locations (15):
- United States (15):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] El-Sadr WM, Manneheimer S, Grant L, Matts J. Use of PCP and MAC prophylaxis among eligible patients with and without CD4+ rebound. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29 (abstract no 129)